CLINICAL TRIAL: NCT04495842
Title: The Effect of Aromatherapy on COVID-19-induced Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nutraceuticals Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20-7-5600
Record Dates: First submitted 2020-07-30; First posted 2020-08-03 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Stress; Covid19; Anxiety
Keywords: aromatherapy; essential oils; environmental health
MeSH Terms: conditions — COVID-19; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants receive an active essential oil blend to inhale for 15 minutes. The blend contains plant based oils sourced from flowers and citrus plants.
  Interventions: Other: Essential Oil Blend
- Control (Placebo Comparator): Participants receive an inert comparison to inhale for 15 minutes.
  Interventions: Other: Control Blend

INTERVENTIONS:
Other: Essential Oil Blend — 5 drops of on a tester strip
  Arms: Intervention
Other: Control Blend — 5 drops on a tester strip
  Arms: Control

SUMMARY:
The purpose of this study is to assess the potential for a non-invasive sensory based intervention to reduce the stress associated with a COVID-19 diagnosis.

DETAILED DESCRIPTION:
After being informed about the study, participants who provide consent will be randomized to one of two groups. Participants will receive one of two aromas to inhale with one being active and the other a control comparison.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy
* Documented COVID-19 exposure, suspected infection, or diagnosed infection
* Has been tested for or diagnosed with COVID-19
* adults age 18-65 living in the US
* understands and agrees to comply with study procedures
* provides informed consent

Exclusion Criteria:

* Smoker in household
* Pregnant or may become pregnant
* Difficulty breathing
* Pain or pressure in the chest
* Confusion
* Hospitalization
* Asthma, COPD, or other respiratory condition
* demonstrated inability to comply with study procedures
* has participated in an interventional clinical study within 31 days prior to enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in state anxiety on the State portion of the State Trait Anxiety Scale (STAI-S) at 15 minutes | Baseline and at 15 minutes
  The STAI-S is a validated self reporting instrument which assesses anxious feelings at that specific moment in time. Possible scores range from 20 to 60, with higher scores pointing to higher anxiety. The STAI-S contains 20 questions which are answered on a Likert scale.
Change from baseline in mood state on the Abbreviated Profile of Mood States (POMS) | Baseline and at 15 minutes
  This instrument contains 40 words such as Lively or Sad, each of which are scored on a scale of 0-4 indicating how much that word refects what they feel in that moment. Scores range from 0-160 with higher scores indicating greater mood disturbances across 7 subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Jessie Hawkins, PhD, Principal Investigator — Nutraceuticals Research Institute
Locations (1):
- Franklin Health Research Center, Franklin, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No